CLINICAL TRIAL: NCT00409851
Title: A 52 Week, Open Label Extension to the Randomized, Double-blind, Multicenter, Multifactorial, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Valsartan and Amlodipine Combined and Alone in Hypertensive Patients.
Brief Title: One Year Study to Evaluate the Safety of the Combination of Valsartan and Amlodipine in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489A2201E1
Record Dates: First submitted 2006-12-07; First posted 2006-12-11 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: HYPERTENSION, VALSARTAN, AMLODIPINE,SAFETY
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan+amlodipine

SUMMARY:
A ONE YEAR SAFETY STUDY FOR PATIENTS WHO COMPLETE STUDY VAA489A2201.

ELIGIBILITY:
Inclusion Criteria:

* SUCCESSFUL COMPLETION OF VAA489A2201 CORE TRIAL
* VISIT 7 BLOOD PRESSURE MUST BE MSDBP ≤ 95 mmHg AND MSSBP ≤ 150 mmHg

Exclusion Criteria:

* PATIENTS WHO EXPERIENCED ANY ADVERSE EVENTS CONSIDERED SERIOUS AND DRUG RELATED IN VAA489A2201 CORE
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1293 (Actual)
Dates: Start 2003-04; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Visit 2) in mean sitting diastolic blood pressure at trough.

SECONDARY OUTCOMES:
Change from baseline (Visit 2) in mean sitting systolic blood pressure at trough
Change from baseline (Visit 2) in standing diastolic and systolic blood pressure at trough
Sitting and standing pulse

CONTACTS AND LOCATIONS:
Overall Officials: Novartis pharmaceuticals, Study Chair — Sponsor GmbH
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Sites in Germany, Germany

REFERENCES:
- See also: NOVARTIS PATIENT RECRUITMENT WEBSITE — http://www.novartisclinicaltrials.com/webapp/etrials/home.do